CLINICAL TRIAL: NCT00996112
Title: Management by Primary Care Clinicians of Patients Suspected of Having Community-Acquired, Methicillin-Resistant Staphylococcus Aureus (CA-MRSA) Infections
Brief Title: Primary Care Management of Community-Acquired, Methicillin-Resistant Staphylococcus Aureus (CA-MRSA) Infections
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Academy of Family Physicians National Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: 09-0265; AHRQ 04-109-6314
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2010-11

CONDITIONS: Methicillin-Resistant Staphylococcus Aureus
Keywords: primary health care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Historical
- Prospective

SUMMARY:
The goal of this study is to further the investigators' understanding of community acquired methicillin-resistant Staph Aureus (CA-MRSA) and treatment of it by developing real-world sustainable strategies consistent with existing guidelines on treatment of CA-MRSA from the Centers for Disease Control and Prevention (CDC) and test these strategies in busy primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting at a primary care clinic who have a skin or soft tissue infection.

Exclusion Criteria:

* None

Max Age: 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises primary care patients in ambulatory clinics from two health care systems.
Sampling Method: Non-Probability Sample
Enrollment: 4518 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Physician Behavior Change | Throughout study participation
  Intervention in practice for guideline-concordant care of CA MRSA

CONTACTS AND LOCATIONS:
Overall Officials: David R West, PhD, Principal Investigator — Department of Family Medicine, University of Colorado Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States